CLINICAL TRIAL: NCT03257800
Title: Laryngeal Mask Insertion Conditions And Hemodynamic Effects After Propofol And Ketamine-Propofol Co-induction
Brief Title: Laryngeal Mask Insertion Conditions And Hemodynamic Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leila mansali stambouli (Other)
Responsible Party: Sponsor-Investigator, Leila mansali stambouli, Principal Investigator and Clinical Professor, University of Monastir
Organization: University of Monastir (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 0925-0586
Record Dates: First submitted 2017-07-16; First posted 2017-08-22 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Laryngeal Masks
Keywords: ketamine; Propofol; laryngeal masks; anesthesia; child
MeSH Terms: interventions — Ketamine; Sevoflurane; Nitrous Oxide

STUDY DESIGN:
Intervention Model Description: Randomized, controlled and double blind assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ketamine-propofol group (Active Comparator): Ketamine (50mg/ml) at 0.5 mg.kg-1 was injected intravenously 1min prior 3 mgkg-1 of propofol and 1 min before LMA insertion in Ketamine-propofol group.
  sevoflurane 6-7% was used on vaporizer setting with 50% nitrous oxide in oxgen prior intravenous anesthesia. The loss of eyelash reflex was considered as the desired end point for induction.
  Interventions: Drug: Ketamine
- propofol group (Placebo Comparator): 0,9% saline solution ( Placebo ) at the same volume as ketamine (50mg/ml) was injected intravenously 1min prior propofol 3 mg.kg-1 and 1 min before LMA insertion in propofol group.
  sevoflurane 6-7% was used on vaporizer setting with 50% nitrous oxide in oxgen prior intravenous anesthesia. The loss of eyelash reflex was considered as the desired end point for induction.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Ketamine — Ketamine 0,5mg.kg-¹was injected intravenously one minute prior propofol 3mg.kg-¹ and one minute before LMA insertion in Ketamine-propofol group
  Other Names: sevoflurane, nitrous oxide (N2O)
  Arms: ketamine-propofol group
Drug: placebo — The control group which received intravenously the same volume with normal saline one minute prior propofol 3mg.kg-¹ and 1 min before LMA insertion in propofol group
  Other Names: sevoflurane, N2O
  Arms: propofol group

SUMMARY:
This interventional double-blind, randomized trial has included120 children of American Society of Anesthesiologist (ASA) physical status I or II aged between 1and 8 years of either sex, scheduled for outpatient minor surgery under general anesthesia.This study examined whether co-induction with ketamine-propofol enhance laryngeal mask airway (LMA) insertion conditions and preserve hemodynamic state in patients.

DETAILED DESCRIPTION:
This study aims to compare two anesthesia protocols: propofol induction with or without a prior injection of ketamine, in term of LMA insertion conditions(favorable= satisfactory or unfavorable= unsatisfactory ) and hemodynamic effects (decrease of 20 % from baseline of blood pressure and heart rate).

The conditions of LMA insertion have been assessed in each study group by an experimented anesthesiologist, who was unaware of the treatment group assignment. Conditions were considered satisfactory, if the 4 following criteria were acceptable: the jaw was relaxed, there was no coughing, swallowing and no limb movement, and then the LMA was inserted. When the investigators save at least one unacceptable of these criteria, conditions were considered to be unsatisfactory and thereafter anesthesia was deepened with supplemental dose of propofol 1mg.kg-¹ and 1 minute later a reinsertion was attempted. The total number of attempts at LMA insertion was recorded. Children trachea was intubated after 3 failed attempts of LMA insertion, and then patient was excluded.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I or II who were scheduled to minor elective ambulatory surgery (e.g. inguinal hernia, undescended testes, umbilical hernia) performed by experienced surgeon under general anesthesia.

Exclusion Criteria:

* patients with full stomach
* A history of gastric reflux
* A history of convulsions, cardiovascular or neuromuscular disease
* Allergies to the study drugs
* obese children
* suspected difficult airway and hyper-reactive airway disease

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2013-12-30 (Actual); Study Completion 2013-12-31 (Actual)

PRIMARY OUTCOMES:
LMA insertion conditions | 2 minutes
  satisfactory conditions of LMA insertion are defined as when 4 criteria were acceptable: jaw relaxation, no coughing or swallowing and no limb movement.
  unsatisfactory conditions of LMA insertion is defined as when there's at least one unacceptable of these criteria

SECONDARY OUTCOMES:
hemodynamic effects | from Baseline period until 10 minutes after LMA insertion
  mean blood pressure (MAP) in mmHg . Heart Rate (HR) in beats per minute (time frame: from baseline to LMA insertion)

OTHER OUTCOMES:
delirium | from awake until 30 min after emergence
  Emergence delirium was assessed by the Pediatric Anesthesia Emergence Delirium Scale (PAED) and was defined as a PAED score >10

CONTACTS AND LOCATIONS:
Overall Officials: leila Mansali Stambouli, MD PhD, Principal Investigator — university Hospital of Fattouma Bourguiba, Monastir, TUNISIA
Locations (1):
- University Hospital of Fattouma Bourguiba, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goel S, Bhardwaj N, Jain K. Efficacy of ketamine and midazolam as co-induction agents with propofol for laryngeal mask insertion in children. Paediatr Anaesth. 2008 Jul;18(7):628-34. doi: 10.1111/j.1460-9592.2008.02563.x. Epub 2008 May 8. PMID 18482245
- [Background] Singh R, Arora M, Vajifdar H. Randomized double-blind comparison of ketamine-propofol and fentanyl-propofol for the insertion of laryngeal mask airway in children. J Anaesthesiol Clin Pharmacol. 2011 Jan;27(1):91-6. PMID 21804715